CLINICAL TRIAL: NCT06299501
Title: How Can Child Health Services Identify and Respond to Family Violence - a Randomized Controlled Trial to Assess the Effectiveness of Routine Questions or Questions Posed on Indication Compared to Treatment as Usual
Brief Title: How Can Child Health Services Identify and Respond to Family Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Jane and Dan Olsson Foundation for Scientific Purposes (Unknown); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lene Lindberg, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LS 2015-1199 and 2017-24
Record Dates: First submitted 2023-12-18; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Family Violence; Domestic Violence; Intimate-partner Violence
Keywords: Family violence; Domestic violence; Intimate-partner violence
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Three-armed study, two intervention groups and one control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine group (Experimental): Nurses within the routine group receive training and are assigned to inform about family violence at the home visit that takes place when the child is newborn and to by routine ask questions about family violence to mothers at the 6-8 weeks visit to CHC.
  Interventions: Procedure: Routine questions
- Indication group (Experimental): Nurses within the indication group receive training and are assigned to inform about family violence at the home visit when the child is newborn and to pose questions about family violence on evidence based indication.
  Interventions: Procedure: Questions on evidence based indication
- Treatment as usual (Active Comparator): Nurses within the treatment as usual group do not receive training but ask questions when they suspect ongoing violence in the family.
  Interventions: Procedure: Treatment as usual

INTERVENTIONS:
Procedure: Routine questions — The routine group of nurses receive training and supervision and will ask questions about family violence to everyone, disregarding if they suspect family violence or not.
  Arms: Routine group
Procedure: Questions on evidence based indication — The group of nurses will receive training and supervision and will ask questions on evidence based indication
  Arms: Indication group
Procedure: Treatment as usual — The group of nurses will ask questions when suspecting ongoing violence in the family
  Arms: Treatment as usual

SUMMARY:
Family violence has severe impacts on children's health and development. The Child Health Services (CHS) in Sweden reaches almost 100% of families with young children and provides a unique setting to facilitate identification of family violence. This study is a three-armed randomized controlled trial (RCT) conducted to assess the effectiveness of different approaches to identify family violence within CHS. Two different approaches are tested and compared to treatment as usual; 1) information about family violence at home visit when child is newborn, and questions posed to all mothers at the 6-8-week visit; 2) information about family violence at home visit when child is newborn, and questions posed to mothers on evidence based indication. Nurses who are randomized into any of the two intervention arms receive training and supervision. The outcomes of the study are related to knowledge, attitudes, and practices around identification and support in case of family violence and number of identified cases of family violence.

DETAILED DESCRIPTION:
Family violence has severe impacts on children's health and development. Early identification of family violence is imperative to facilitate timely interventions. In Sweden, the Child Health Services (CHS) has a main aim to promote children's health and development and prevent ill health. The Swedish CHS program reaches almost 100% of families and includes 18 scheduled visits characterized by a health-promoting approach focusing on the child and the parents' wellbeing. The CHS offers a unique setting to identify family violence among families with young children. However, there is a paucity of knowledge on how questions about family violence should be addressed within CHS. The aim of the study is to increase knowledge of the effectiveness of an evidence-based program within the Swedish CHS to identify family violence. The specific research question is: How can practice within CHS contribute to identification of family violence on routine or indication compared to treatment as usual?

A three-armed pragmatic randomized controlled trial (RCT) was conducted in 2017-2019 where all CHS's (n=120) in Region Stockholm were invited to participate. A total of 85 nurses from 22 CHC's participated in the trial of which 32 nurses from 10 CHS's were assigned the routine arm, 25 nurses from 5 CHS's were assigned the evidence based indication arm and 28 nurses from 7 CHS's were assigned to the treatment as usual group. Randomization was performed on CHS level so that the same approach was followed at each CHS when the first nurse was randomized. Only nurses in the routine and indication groups received training and supervision. The group that was assigned treatment as usual was offered the same training after the study was completed. The nurses completed questionnaires on the outcome knowledge, attitudes, and practices to identify and deal with family violence at three time points. Nurses in the two intervention groups also documented their practices and any identified cases of family violence during the intervention.

The findings of the study can contribute to knowledge on how children exposed to family violence can be identified and adequate measures be put in place.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurse
* Working in any of the Child Health Services in the Stockholm Region

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitudes and practices | Measured before randomization, within two weeks after training and six months post-training.
  An adaptation of the "Physician Readiness to Manage Violence Survey" developed by Short LM et al. (Am J Prev Med 2006; 30(2):173-180) and Ramsay J et al. (Brit J Gen Pract 2012; 62(602):647-655) was used. Higher values indicate more positive outcomes.
  A subscale was used to measure knowledge about definition, prevalence and consequences of family violence (FV), summarized into a total value, with higher values indicating higher knowledge. Additional questions concerned knowledge of guidelines, reporting to social services and local interventions for children and parents.
  Nurse's attitudes by asking about informing, asking questions about and acting upon FV.
  Practices were measured by questions about how nurses provided or displayed information material, asked about FV and their reports of concern to social services.

SECONDARY OUTCOMES:
Number of cases of family violence | Documentation covers the intervention phase (6 months)
  Documentation from nurses in the two intervention arms on number of identified cases of family violence

CONTACTS AND LOCATIONS:
Overall Officials: Lene Lindberg, Principal Investigator — Karolinska Institutet
Locations (1):
- Central Child Health Care (Centrala barnhälsovården), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No